CLINICAL TRIAL: NCT03130517
Title: Efficacy of Intravenous Immunoglobulin in Management of RH and ABO Incompatibility Disease of Newborn and Its Effect in Decrease Duration of Hospital Stay and Need for Exchange Transfusion
Brief Title: Efficacy of Intravenous Immunoglobulin in Management of Rh and ABO Incompatibility Disease
Acronym: IVIG
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem ahmed, Doctor, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: assuit university 66
Record Dates: First submitted 2017-04-24; First posted 2017-04-26 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Haemolysis Neonatal
Keywords: hemolysis,newborn
MeSH Terms: conditions — Hemolysis | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: intervention group will recieve intravenous immunoglobulin and phototherapy and control group that will receive phototherapy only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Other): Use of single dose of intravenous immunoglobulin in a dose 0.5_1gm /kg to intervention group
  Interventions: Drug: intravenous immunoglobulin
- Control group (Other): Control group will recieve phototherapy only
  Interventions: Drug: intravenous immunoglobulin

INTERVENTIONS:
Drug: intravenous immunoglobulin — giving intravenous immunoglobulin to neonates included in inclusion criteria in a dose of 0.5-1 gm
  Other Names: gammaglobulin

SUMMARY:
hemolytic disease of newborn is an important cause of hyperbilirubinemia with significant morbidity and mortality in neonatal period. intravenous immunoglobulin has widely used in management of hemolytic disease of new born

DETAILED DESCRIPTION:
Hemolytic disease of the newborn (HDN) due to red cell alloimmunisation is an important cause of hyperbilirubinemia with significant morbidity in the neonatal period . Hemolytic disease of the newborn has unfortunately continued to contribute to perinatal and neonatal morbidity and mortality in developing countries . The degree to which the fetus is affected correlated with the amount of maternal antibody that cross the placenta .

Hemolysis from ABO incompatibility is one of the most common cause of isoimmune hemolytic disease during neonatal period. Infants with blood group type A or B , carried by blood group type O mother, will have a positive antibody because of maternal anti-A or anti-B transfer in to the fetal circulation. Ten percent of these infants will present with hemolytic disease . Most of the infant presents with unconjugated hyperbilirubinemia in the first 24 h of life and it is rarely a cause in patients who are discharged from nursery and readmit with severe hyperbilirubinemia.

Rh incompatibility can occur when an Rh-negative pregnant mother is exposed to Rh-positive fetal red blood cells secondary to fetomaternal hemorrhage during the course of pregnancy from spontaneous or induced abortion , trauma, invasive obstetric procedures, or normal delivery. As a consequence, blood from the fetal circulation, and, after a significant exposure, sensitization occurs leading to maternal antibody production against the foreign Rh antigen. Once produced, maternal Rh immunoglobulin G (IgG) antibodies may cross freely from the placenta to the fetal circulation, where they form antigen-antibody complexes with Rh- positive fetal erythrocytes and eventually are destroyed, resulting in a fetal alloimmune-induced hemolytic anemia and Jaundice.

Traditional neonatal treatment of HDN consists of intensive phototherapy and exchange transfusion (ET). However, ET is a high-risk invasive procedure associated with a significant rate of adverse effects .Although the mortality rate associated with ET is currently reported to be less than 0.3% in term infants , the morbidity rates can reach 74% and includes catheter-related complications, sepsis, thrombocytopenia and hypocalcemia

Intravenous Immunoglobulin G (IVIG) therapy has been widely used for a variety of indications in newborn period such as alloimmune neonatal thrombocytopenia and an adjunctive treatment of neonatal infections. American Academy of Pediatrics, recommends high dose IVIG (0.5_1 g/kg) as an additional treatment of Rh and ABO hemolytic disease and its use however there is no consensus on its routine use in ABO hemolytic disease yet .

IVIG "contains a spectrum of antibodies capable of interacting with and altering the activity of cells of the immune system as well as antibodies capable of reacting with cells such as erythrocytes". When hemolytic disease occurs, maternal antibodies present in the infant's blood attach to the antigen receptors on the infant's red blood cells. Specifically, the maternal antibody attaches its Fc region, the lower portion of the antigen, to specific immune system cells , such as machrophages, stimulating the destruction of the antigen-antibody complex and the red blood cell. It has been proposed that IVIG blocks the Fc receptor and therefore blocks the binding of the antibody to the antigen. With this blockade, hemolysis no longer occurs.

Neonatal treatment with intravenous immunoglobulin (IVIG) has been suggested as an altenative therapy to ET for isoimmune hemolytic jaundice to reduce the need for exchange transfusion and duration of phototherapy and hospitalization in isoimmune hemolytic disease of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* 1)Gestational age more than or equal 37 weeks and postnatal age from 48hr-72hr.

  2)Anemia with Reticulocytic count 10% 3)Serum total bilirubin around 18mg/dl .

Exclusion Criteria:

* 1)perinatal asphyxia. 2)Congenital malformation. 3)Severe respiratory distress. 4)Sepsis during hospital stay. 5)Metabolic problems . 6)Gestational age less than 37 weeks

Ages: 48 Hours to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure duration of phototherapy | Two days
  to measure how many neonate need for exchange transfusion after one dose of intravenous immunoglobulin and reduction of haemolysis rate which is estimated by reduction in reticulocytic count

SECONDARY OUTCOMES:
duration of hospital stay | Four days
  neonates with intravenous immunoglobulin is expected to stay less in hospital and decrease duration of phototherapy

IPD SHARING:
Plan to Share IPD: Undecided
patients with Rh and ABO incompatibility disease will recieve intravenous immunoglobulin